CLINICAL TRIAL: NCT05043389
Title: Impact of Myofuntional Therapy Program on Increasing Tongue Strength and Improving Sleep Apnea: a Randomized Controlled Trail
Brief Title: Impact of Myofuntional Therapy Program on Increasing Tongue Strength and Improving Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 63238
Record Dates: First submitted 2021-09-05; First posted 2021-09-14 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2021-09

CONDITIONS: Obstructive Sleep Apnea
Keywords: myofunctional therapy; IOPI; Obstructive sleep apnea (OSA)
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Obstructive sleep apnea (Experimental): myofunctional therapy program
  Interventions: Other: myofunctional therapy program
- control (No Intervention): standard treatment

INTERVENTIONS:
Other: myofunctional therapy program — Exercise oral cavity muscle
  Arms: Obstructive sleep apnea

SUMMARY:
This Research studies for compare muscle strength among OSA patients who treat with myofunctional therapy program in Rajavithi hospital

ELIGIBILITY:
Inclusion Criteria:

* Patients who diagnose with Obstructive sleep apnea 18-65 years

Exclusion Criteria:

* BMI>=35kg/m2
* alcoholic and smoke
* use sleeping pill
* craniofacial syndrome
* hypertrophic tonsils grade 3+, 4+
* severe comorbidity
* Use CAP

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Compare muscle strength | 1 year
  compare muscle strength before and after program by IOPI

CONTACTS AND LOCATIONS:
Overall Officials: Sasion Phaibunphunphiphat, MD, Principal Investigator — Department of Medical Services Ministry of Public Health of Thailand
Locations (1):
- Rajavithi Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided